CLINICAL TRIAL: NCT02658396
Title: A Phase I Trial of the MUC1 Inhibitor, GO-203-2c, in Combination With Bortezomib in Patients With Relapsed or Refractory Multiple Myeloma
Brief Title: GO-203-2C + Bortezomib For Relapsed Or Refractory MM
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study was never open due to lack of funding
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Genus Oncology, LLC (Industry); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Jacalyn Rosenblatt, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-363
Record Dates: First submitted 2016-01-13; First posted 2016-01-18 (Estimated); Last update posted 2017-07-05 (Actual); Status verified 2017-06

CONDITIONS: Multiple Myeloma; Multiple Myeloma in Relapse; Refractory Multiple Myeloma
Keywords: Multiple Myeloma; Relapsed Multiple Myeloma; Refractory Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- GO-203-2C (Experimental): * Patients who fulfill eligibility criteria will be entered into the trial to receive Bortezomib and GO-203-2C.
  * After the screening procedures confirm participation in the research study:
  The investigators are looking for the highest dose of the combination of study drugs that can be administered safely without severe or unmanageable side effects in participants that have multiple myeloma, not everyone who participates in this research study will receive the same dose of the study drug. The dose given will depend on the number of participants who have been enrolled in the study prior and how well the dose was tolerated.
  * Bortezomib
  * GO-203-2C
  Interventions: Drug: GO-203-2C; Drug: Bortezomib

INTERVENTIONS:
Drug: GO-203-2C
Drug: Bortezomib
  Other Names: Velcade

SUMMARY:
This research study is studying a combination of targeted therapies known as GO-203-2C and bortezomib as a possible treatment for multiple myeloma that has either progressed or not responded to treatment.

DETAILED DESCRIPTION:
This research study is a Phase I clinical trial, which tests the safety of an investigational intervention and also tries to define the appropriate dose of the investigational intervention to use for further studies. "Investigational" means that the intervention is being studied.

The FDA (the U.S. Food and Drug Administration) has not approved GO-203-2C as a treatment for any disease.

The FDA (the U.S. Food and Drug Administration) has approved bortezomib as a treatment option for your disease.

The purpose of this research study is to test the safety of GO-203-2C with bortezomib. GO-203-2C is a newly discovered compound that binds to an oncoprotein (a cancer causing protein) called MUC1. Myeloma cells harbor an increased amount of MUC1 on its cell surface. By binding to MUC1, GO-203-2C has been shown to cause tumor cell death in laboratory studies.

Bortezomib is an intravenously or subcutaneously administered medication that belongs to a class of drugs called proteasome inhibitors. Proteasome inhibitors disrupt the normal action of cells that breakdown proteins in both normal and cancer cells. This disruption can stall tumor growth and cause cancer cells to die. Bortezomib is currently approved for the treatment of multiple myeloma.

The Investigators want to find the highest dose of GO-203-2C given in combination with bortezomib that can be administered safely without severe or unmanageable side effects.

ELIGIBILITY:
Inclusion Criteria:

* Participants with multiple myeloma who experienced disease progression after the most recent treatment regimen. Patients must have had prior treatment with a proteasome inhibitor, immunomodulatory drug, and if eligible for transplant an autologous transplant.
* Patients must have measurable disease, defined as 1 or more of the following:

  * serum M-protein > 0.5 g/dL. For patients with IgA myeloma where the M-protein cannot be quantified on SPEP, total IgA > 0.5 g/dL.
  * Urine M-protein > 200mg/24h
  * serum FLC assay: involved FLC level > 10 mg/dL with abnormal FLC ratio
* Greater than or equal to 18 years in age
* ECOG performance status ≤2 (see Appendix A)
* Life expectancy of greater than 3 months
* Participants must have normal organ and marrow function as defined below:

  * leukocytes ≥2,000/mcL
  * platelets ≥50,000/mcL
  * total bilirubin ≤ 2.0 mg/dL (patients with Gilbert syndrome and Bilirubin ≤ 3.5 mg/dL are eligible)
  * AST(SGOT)/ALT(SGPT) ≤2.5 × institutional upper limit of normal
  * creatinine ≤ 2 mg/dL

    --- OR
  * creatinine clearance ≥60 mL/min/1.73 m2 for participants with creatinine levels above institutional normal.
* Women of child-bearing potential must have a documented negative pregnancy test.
* The effects of GO-203-2c on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of GO-203-2c administration.
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Participants who have had chemotherapy or radiotherapy within 14 days (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 14 days earlier. The use of steroids up the equivalent of 160 mg of dexamethasone is allowed within 14 days of screening, but the last dose has to be given at least 1 day prior to initiation of treatment.
* Participants who are receiving any other investigational agents.
* Uncontrolled hypertension. This is defined as sustained blood pressure elevation > 140/90 despite antihypertensive therapy. Patients are allowed to start antihypertensive therapy to meet eligibility criteria; however they have to be on a stable antihypertensive regimen for at least 7 days.
* Uncontrolled intercurrent illness including, but not limited to, uncontrolled infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because GO-203-2c is an agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with GO_203-2c, breastfeeding should be discontinued if the mother is treated with GO-203-2c. These potential risks may also apply to other agents used in this study.
* Individuals with a history of a different malignancy are ineligible except for the following circumstances: Individuals with a history of other malignancies are eligible if they have been disease-free for at least 5 years and are deemed by the investigator to be at low risk for recurrence of that malignancy. Individuals with the following cancers are eligible if diagnosed and treated within the past 5 years: cervical cancer in situ, and basal cell or squamous cell carcinoma of the skin.
* Hypersensitivity to bortezomib, boron or mannitol.
* Grade 3 or 4 peripheral neuropathy.
* Prior discontinuation of a bortezomib-based therapy due to toxicity attributed to bortezomib.
* Use of G-CSF administration within 7 days of screening
* Platelet transfusion within 7 days of screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2019-05 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
MTD Dose | Baseline to 21 Days

SECONDARY OUTCOMES:
Response Rate | 12 Months
Progression Free Survival | Start of treatment to disease progression or death from any cause, assessed up to 100 months
  Estimated using the method of Kaplan and Meier.
Event Free Survival | Time of treatment initiation to Progressive Disease, death, or nonprotocol therapy, assessed up to 100 months
  Estimated using the method of Kaplan and Meier.
Time-to-new treatment | From treatment initiation to next treatment or death of any cause, assessed up to 100 months
  Estimated using the method of Kaplan and Meier.

CONTACTS AND LOCATIONS:
Overall Officials: Jacalyn Rosenblatt, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (2):
- United States (2):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts